CLINICAL TRIAL: NCT05927493
Title: Analysis of the Outcome of Patients With Suspected Upper GI Bleeding Managed in Emergency Departments in Ile de France and External Validation of Prognostic Scores
Brief Title: Patients With Upper Gastrointestinal Bleeding in Emergency Department
Acronym: UGIB-ED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0034
Record Dates: First submitted 2023-05-11; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Upper gastrointestinal bleeding; Emergency department; Low-risk; Scores
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Upper gastrointestinal bleeding: Patients with upper gastrointestinal bleeding hospitalized after ED visit

SUMMARY:
More than 80% of patients with upper gastrointestinal bleeding (UGIB) are hospitalized after their visit to the emergency department (ED). However, some of these hospitalizations do not seem justified. Several clinical scores have been developed to classify patients according to their risk of death or need for therapeutic intervention.

The aims of this study are:

1. to describe the characteristics of patients hospitalized for UGIB after their visit to the ED
2. to assess the predictive factors of hospital intervention or death
3. to assess the accuracy of existing prognostic scores to classify patients according their risk of death or need for therapeutic intervention (external validation) and to identify low-risk patients not requiring intervention.
4. Depending on the results, a new score could be derived to identify patients at low risk for intervention or death.

DETAILED DESCRIPTION:
Upper gastrointestinal bleeding (UGIB) is caused by several conditions, with an overall mortality of approximately 10%. More than 80% of patients are hospitalized after their visit to the emergency department (ED) [1]. The hospitalization usually allows an etiological diagnosis to be made by performing an upper gastrointestinal endoscopy (UGE) and a hemostatic treatment if required. However, some of these hospitalizations do not seem justified. Indeed, some patients do not require any intervention (i.e., blood transfusion, endoscopic, radiological or surgical hemostasis) and have no complications (i.e., rebleeding, death). Some of them do not even have a diagnostic UGE during their hospital stay.

Several clinical scores have been developed to classify patients according their risk of death or need for therapeutic intervention, some of them to identify patients with low-risk of complications (rebleeding, death) and/or need for intervention. The most commonly known are the pre-endoscopic Rockall score, the Glasgow-Blatchford Score (GBS) and the AIMS65. Among them, the GBS seems to be the most efficient [2,3]. Its use is encouraged in the latest French, European and international recommendations [4].

Other prognostic scores have more recently been proposed with this purpose (e.g. modified GBS, CANUKA, H3B2, C-Watch, Harbinger), with interesting results but scarce or no external validation.

The aims of this study are:

1. to describe the characteristics of patients hospitalized for UGIB after their visit to the ED
2. to assess the predictive factors of death or therapeutic intervention (i.e, blood transfusion, endoscopic hemostasis, surgery or interventional radiology)
3. to assess the accuracy of existing prognostic scores to classify patients according their risk of death or need for therapeutic intervention (external validation) and to identify low-risk patients not requiring intervention.
4. Depending on the results, a new score could be derived to identify patients at low risk for intervention or death.

ELIGIBILITY:
Inclusion Criteria:

* patient ≥ 18 years old
* with a diagnosis of upper gastrointestinal bleeding (defined by ICD10 codes)
* visited a hospital with ED data available in the data warehouse

Exclusion Criteria:

* reason for consultation not related to upper gastrointestinal bleeding (identified by manual reading of hospital notes)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient ≥ 18 years old with a diagnosis of upper gastrointestinal bleeding hospitalized after an ED visit in hospital with data available in the Assistance Publique-Hôpitaux de Paris data warehouse
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Number of patients treated with specific therapeutic intervention | 7 days
  Blood transfusion or endoscopic hemostasis or radiological hemostasis or surgical hemostasis in 7 days
Number of deceased patients | 30 days

SECONDARY OUTCOMES:
Number of patients treated with blood transfusion(s) | 7 days
  Transfusion of at least 1 red blood cell unit
Number of patients treated with endoscopic hemostasis | 7 days
  Any hemostasis technique used during upper gastrointestinal endoscopy
number of patients treated with endoscopic hemostasis | 7 days
  Arterioembolization or transjugular intrahepatic portosystemic shunt placement
number of patients treated with interventional radiology hemostasis | 7 days
  Any hemostasis technique used during surgery
Death | 30 days
  Intrahospital death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Clément THIEBAUD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency department:Saint-Antoine Hospital, Paris, France